CLINICAL TRIAL: NCT07133516
Title: A Multi-center Study on Artificial Intelligence-Based Quantitative Evaluation of Echocardiography
Acronym: MAIQUEE
Status: Recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Chief of Cardiovascular Ultrasound, First Hospital of China Medical University
Other Study IDs: MAIQUEE STUDY
Record Dates: First submitted 2025-07-30; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Artificial Intelligence (AI); Artificial Intelligence (AI) in Diagnosis; Cardiovascular Diseases (CVD); Echocardiography
Keywords: Artificial Intelligence (AI); Artificial Intelligence (AI) in Diagnosis; Cardiovascular Diseases (CVD); Echocardiography
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AI group: The cardiac chamber size and functional parameters of all 1600 subjects were measured by AI
- Senior physician group: The cardiac chamber size and functional parameters of all 1600 subjects were measured by senior physicians at the PI unit
- Intermediate physician group: The cardiac chamber size and functional parameters of all 1600 subjects were measured by intermediate physicians at each sub center

SUMMARY:
This project aims to collaborate with multiple medical institutions to verify the accuracy, stability, and clinical application value of AI algorithms in echocardiographic quantitative measurement through multi-center clinical research. Specific objectives include:

1. Compare the automatic measurement results of AI with the manual measurement data from physicians of different levels, and analyze the measurement deviation and consistency of AI in key parameters such as intracardiac diameter, volume, and function.
2. Investigate whether AI-assisted measurement can significantly reduce echocardiogram analysis time and optimize clinical workflows. Through multi-center data validation, establish a standardized reference system for AI ultrasound measurement, promote the promotion and application of AI technology in medical institutions at all levels, and reduce diagnostic differences between different hospitals and physicians.
3. Exploring the application of AI in special cases: Assessing the measurement stability of AI algorithms in complex cases (such as cardiomyopathy, valvular disease, coronary heart disease, etc.), and optimizing AI models to meet broader clinical needs.

DETAILED DESCRIPTION:
Cardiovascular disease is a major threat to the health of Chinese residents, and echocardiography, as its core diagnostic tool, directly affects clinical decision-making in terms of measurement accuracy and efficiency. However, traditional ultrasound evaluation heavily relies on physician experience, with pain points such as strong subjectivity, time-consuming measurements, and uneven levels of primary diagnosis. There is an urgent need for technological innovation to improve diagnostic standardization. In recent years, artificial intelligence (AI) technology has shown great potential in the field of medical image analysis, which can achieve automated quantitative measurement of cardiac chamber structure and function. However, existing AI models generally have problems such as insufficient multi center validation and limited adaptability to complex cases, which restrict their clinical translation and application.

To overcome these bottlenecks, this project collaborates with multiple medical institutions to conduct clinical research, systematically evaluating the measurement differences between AI algorithms and physicians of different levels, and assessing the accuracy and stability of AI algorithms. The research will focus on verifying the value of AI technology in improving diagnostic consistency, optimizing workflows, and exploring its potential applications in complex cardiovascular diseases. By establishing a standardized evaluation system, this project aims to promote the standardized application of AI ultrasound technology, ultimately achieving the goal of improving diagnosis and treatment efficiency, promoting the sinking of high-quality medical resources, and helping to improve the overall level of cardiovascular disease prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 - 80 years;
2. Types of diseases (8 in total, 200 cases each):

   1. Normal heart
   2. Coronary heart disease (with segmental thinning and abnormal movement)
   3. Valve disease (valve stenosis or reflux)
   4. Hypertensive heart disease
   5. Atrial fibrillation
   6. Heart failure
   7. Dilated cardiomyopathy
   8. Hypertrophic cardiomyopathy

Exclusion Criteria:

1. Patients with congenital heart disease
2. Patients with poor image quality

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who require cardiac ultrasound examination for various reasons in clinical practice. Ultrasound and clinical diagnosis of patients with normal cardiac structure and function, as well as those with coronary heart disease, valve disease, hypertensive heart disease, atrial fibrillation, heart failure, dilated cardiomyopathy, and hypertrophic cardiomyopathy. A total of 1600 adults were enrolled in multiple centers;
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The indicators of left ventricular size and function are measured by AI, senior physicians at the PI unit, and intermediate physicians at each sub center respectively (all parameters are measured by Mindray ultrasonic machines on the machine) | Artificial intelligence and intermediate doctors measurement results of each sub center will be completed within one day after data collection. Senior physicians measurement results of PI unit will be completed within one month after data collection.
  Left ventricular end diastolic volume (EDV, ml), end systolic volume (ESV, ml), and ejection fraction (EF, %) (calculated by (EDV-ESV)/EDV*100% ) in the four chamber view and two chamber view, as well as the Simpson biplane left ventricular volume (ml) and ejection fraction (%) results.
The indicator of right ventricular function is measured by AI, senior physicians at the PI unit, and intermediate physicians at each sub center respectively (all parameters are measured by Mindray ultrasonic machines on the machine) | Artificial intelligence and intermediate doctors measurement results of each sub center will be completed within one day after data collection. Senior physicians measurement results of PI unit will be completed within one month after data collection.
  Right ventricular area change rate calculated by (EDA-ESA)/EDA*100%.
The indicators of right ventricular size are measured by AI, senior physicians at the PI unit, and intermediate physicians at each sub center respectively (all parameters are measured by Mindray ultrasonic machines on the machine) | Artificial intelligence and intermediate doctors measurement results of each sub center will be completed within one day after data collection. Senior physicians measurement results of PI unit will be completed within one month after data collection.
  Right ventricular end diastolic area (EDA) and end systolic area (ESA).

SECONDARY OUTCOMES:
Doppler ultrasound measurement indicators by are measured by AI, senior physicians at the PI unit, and intermediate physicians at each sub center respectively (all parameters are measured by Mindray ultrasonic machines on the machine) | Artificial intelligence and intermediate doctors measurement results of each sub center will be completed within one day after data collection. Senior physicians measurement results of PI unit will be completed within one month after data collection.
  Forward blood flow velocity of mitral and tricuspid valve (m/s).
Mitral valve annulus and tricuspid valve annulus displacement are measured by AI, senior physicians at the PI unit, and intermediate physicians at each sub center respectively (all parameters are measured by Mindray ultrasonic machines on the machine) | Artificial intelligence and intermediate doctors measurement results of each sub center will be completed within one day after data collection. Senior physicians measurement results of PI unit will be completed within one month after data collection.
  Mitral valve annulus and tricuspid valve annulus displacement (mm)

CONTACTS AND LOCATIONS:
Locations (37):
- China (37):
  - Huainan First People's Hospital, Huainan, Anhui
  - Union Hospital Affiliated to Fujian Medical University, Fuzhou, Fujian
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - Shenzhen Hospital of Fuwai Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Youjiang Medical University for Nationalities, Baise City, Guangxi
  - Guilin Hospital of Traditional Chinese Medicine, Guilin, Guangxi
  - The Fourth Affiliated Hospital of Guangxi Medical University / Liuzhou Workers' Hospital, Liuchow, Guangxi
  - Yulin First People's Hospital, Yulin, Guangxi
  - The Second Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Haikou People's Hospital, Haikou, Hainan
  - The Second Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Loudi First People's Hospital, Loudi, Hunan
  - Hunan Province Directly Affiliated TCM Hospital, Zhuzhou, Hunan
  - Baotou No.4 Hospital, Baotou, Inner Mongolia
  - Shangrao Central Hospital, Shangrao, Jiangxi
  - Shangrao People's Hospital, Shangrao, Jiangxi
  - Ansteel Group General Hospital, Anshan, Liaoning
  - Chaoyang Central Hospital, Chaoyang, Liaoning
  - Fushun Central Hospital, Fushun, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qinghai Provincial Hospital of Cardiovascular and Cerebrovascular Diseases, Xining, Qinghai
  - The Central Hospital Affiliated to Shandong First Medical University, Tai’an, Shandong
  - Linfen People's Hospital, Linfen, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Jiangyou 903 Hospital, Jiangyou, Sichuan
  - Bishan Hospital Affiliated to Chongqing Medical University, Chongqing
  - Bishan Hospital Affiliated to Chongqing University of Chinese Medicine (Chongqing Bishan District Hospital of Traditional Chinese Medicine), Chongqing
  - Chongqing Hospital of Traditional Chinese Medicine, Chongqing
  - Chongqing People's Hospital, Chongqing
  - Fuling Hospital Affiliated to Chongqing University, Chongqing
  - The First Affiliated Hospital of Army Medical University, Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Shanghai Changzheng Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided